CLINICAL TRIAL: NCT04200209
Title: The Implementation and Impact of a Rapid-cycle Quality Indicator Feedback Mechanism on Patients and Professionals: a Case Study of Sint-Trudo Hospital
Brief Title: To a Sustainable Quality Policy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Sint-Trudo Hospital (Other)
Responsible Party: Principal Investigator, Kris Vanhaecht, Professor, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SQP4ST
Record Dates: First submitted 2019-12-11; First posted 2019-12-16 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Quality Improvement; Public Health; Management Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hospital (Experimental): Twelve wards of the hospital will be evaluated at the same time.
  Interventions: Other: Implementation of a quality indicator feedback mechanism

INTERVENTIONS:
Other: Implementation of a quality indicator feedback mechanism — 1. Audit and feedback: A summary of clinical performance and hospital safety culture over a specified period of time.
  2. Benchmarking Achievable: benchmarks are calculated from the performance of all members of a peer group and represents a realistic standard of excellence attained by the top performers in that group (i.e. comparing to the top 10% of peers).
  3. Educational outreach: A trained independent person or investigator will meet with health professionals or managers in their practice setting to provide information (e.g. feedback of quality indicators).
  4. Action planning: The purpose of action planning is to support quality improvement efforts by identifying opportunities for improvement, strategies and steps to accomplish the work.

SUMMARY:
The investigators need stronger feedback loops and a quality monitoring and management system to improve the quality of care in sustainable way. The Chair Sint-Trudo "To a sustainable quality policy" was established to scientifically develop prerequisites for a sustainable quality of care. In this study protocol, a monocentric mixed-method quasi-experimental study will be used to assess the impact of a rapid-cycle quality indicator feedback mechanism on both patients and professionals.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in the hospital for more than one night

Exclusion Criteria:

* Patients admitted in the hospital for less than one night

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Hospital mortality | During admission
  In-hospital mortality rate
Patient experiences | During admission
  Experiences of patients will be measures by a validated questionnaire (Flemisch Patient Experience Questionnaire).
  Q: Will you recommend our hospital? (scale min 0 until 10 with 0: not and 10: for sure).
  For follow questions the scores are 'disagree', 'somewhat agree', 'largely agree', 'totally agree. The higher the score the better the outcome Q: This information was provided by my GP or by healthcare providers in the hospital.
  Q: I understand the information I received about the cost of my stay. Q: I received sufficient information about the causes of my condition or about the possible treatment methods for my condition or about the consequences of my disease.
  Q: Nurses or doctors explained things in a way I could understand or treated me with courtesy and respect.
  Q: My privacy was respected during conversations with caregivers or during examinations, treatment and care.
  Q: Before any treatment my identity was checked. Q: Hospital staff always introduced themselves
In-hospital length of stay | During admission
  Length of stay of each patient in the hospital
Adverse events and adverse outcomes | During admission
  Each adverse event and following adverse outcomes will be measured: urinary tract infections, pressure ulcers, hospital-acquired pneumonia, shock/cardiac arrest, upper-gastrointestinal bleeding, hospital-acquired sepsis, deep venous thrombosis, central nervous system complications, surgical wound infection, pulmonary failure, metabolic derangement, methicillin-resistant Staphylococcus aureus, vancomycin resistant Enterococcus, central line associated bloodstream infections, carbapenemase producing Enterobacteriaceae
Failure to rescue rate | During admission
  The failure to rescue rate for each patient admitted in the hospital will be evaluated
Readmission rate | 30 days after discharge
  Readmission within 30 days of each patient admitted in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Kris Vanhaecht, MSc, Principal Investigator — Professor
Locations (1):
- Sint-Trudo Ziekenhuis, Sint-Truiden, Belgium